CLINICAL TRIAL: NCT05877300
Title: Safety and Feasibility Study of the CELLSPAN Esophageal Implant (CEI) in Patients Requiring Short Segment Esophageal Replacement
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Harvard Apparatus Regenerative Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSTG-CEI-101
Record Dates: First submitted 2023-05-05; First posted 2023-05-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Diseases
Keywords: Esophagus; Esophagectomy; Tissue Engineering; Organ Regeneration; Regenerative Medicine; Cell Therapy; Dual Arm; Unblinded; Multicenter; FIH; CEI
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Short Segment Esophageal Replacement in patients requiring a full reconstruction of the esophagus (Experimental)
  Interventions: Combination Product: CEI Thoracic Surgical Implantation-Cellspan™ Esophageal Implant-Adult (CEI) in patients requiring a full reconstruction of the esophagus
- Short Segment Esophageal Replacement in patients that have had a previous partial esophagectomy (Experimental)
  Interventions: Combination Product: CEI Extra-Thoracic Subdermal Surgical Implantation - Cellspan™ Esophageal Implant-Adult (CEI) in patients that have had a previous partial esophagectomy

INTERVENTIONS:
Combination Product: CEI Thoracic Surgical Implantation-Cellspan™ Esophageal Implant-Adult (CEI) in patients requiring a full reconstruction of the esophagus — The CEI will be surgically implanted using standard thoracotomy techniques for esophageal reconstruction. Day 0 procedures include: a short segment esophageal resection up to 6 cm, CEI implantation with end-to-end anastomosis, placement of a covered metallic stent, securing the stent with sutures, measuring and recording the stent position, placing draining catheters, inserting a dual lumen gastric-jejunal feeding tube, and conducting hematology and serum tests. A baseline CT/MRI scan will be performed post-surgery to check the anastomotic sites and stent placement.
  Arms: Short Segment Esophageal Replacement in patients requiring a full reconstruction of the esophagus
Combination Product: CEI Extra-Thoracic Subdermal Surgical Implantation - Cellspan™ Esophageal Implant-Adult (CEI) in patients that have had a previous partial esophagectomy — For CEI grafts extending the upper esophagus from the neck ostomy, the patient is positioned supine to expose the left neck and upper chest. A neck incision is made medial to the sternocleidomastoid muscle. The distal esophagus at the cervical spit fistula is freed and mobilized. The CEI is connected to the mobilized esophageal segment with absorbable sutures. Photos document the new spit fistula length post-graft. A new spit fistula tunnel is created on the anterior chest wall, preserving skin and tissue. A covered metallic stent is placed endoscopically through the spit fistula into the CEI, secured with sutures. Pre-surgery tests include hematology, serum chemistry, urinalysis, and CRP, with CRP checked on Days 3 and 5 post-surgery. A CT or MRI scan is done on days 3-7 post-surgery to establish a baseline for tissue deposition analysis around the CEI.
  Arms: Short Segment Esophageal Replacement in patients that have had a previous partial esophagectomy

SUMMARY:
Cellspan™ Esophageal Implant-Adult (CEI)

The CEI is a combination product consisting of an engineered synthetic scaffold (device constituent) seeded and cultured with the patient's adipose derived mesenchymal stem cells (biologic constituent), intended to stimulate regeneration of a structurally intact, living biologic esophageal conduit, in patients requiring full circumferential esophageal reconstruction up to 6 cm segment in length.

This is a dual arm, unblinded, multicenter, prospective first-in-human (FIH) feasibility study to be performed at a maximum of 5 centers in the United States with a maximum of 10 subjects in total. All subjects will be followed for a minimum of 2 years post-implant surgery.

Since this is an FIH experience, the study will utilize an independent Data Monitoring Committee (DMC) to evaluate safety on a continuous basis to mitigate any safety risks to subjects. A sentinel approach to enrollment of subjects shall be guided by the DMC review of cases.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

1. Subject ≥18 years of age
2. The patient has medical conditions requiring esophageal reconstruction, such as, but not limited to:

   1. Refractory benign esophageal strictures (RBES)
   2. Esophageal perforation (full thickness)
   3. Chronic/persistent esophageal fistula
   4. Combination of esophageal perforations/fistula with RBES
3. The patient must have failed at least 3 previous treatment modalities to correct the medical esophageal condition (a-d).

   a. If RBES: i. Steroid treatment ii. Esophageal balloon dilation (EBD) iii. Stent use ≥ 6 months iv. Endoscopic incisional repair

   b. If esophageal perforation: i. Fibrin glue ii. Endoscopic clips and/or suturing iii. Stent use ≥ 6 months iv. Primary surgical repair

   c. If Chronic/Persistent fistula(e): i. Fibrin glue ii. Endoscopic clips and/or suturing iii. Stent ≥ 6 months iv. Primary surgical repair

   d. If Combination Perforation/fistula with RBES i. Fibrin glue ii. Endoscopic clips and/or suturing iii. Stent use ≥ 6 months iv. Primary surgical repair
4. The patient must be a surgical candidate for a short segment esophageal reconstruction (≤6 cm full circumferential segmental excision)
5. The location of the esophageal segment for surgical resection is within the thoracic cavity, defined as, above the diaphragm and at least 4 cm below the larynx.
6. The patient must be a high-risk candidate for minimally invasive esophageal reconstruction, based upon the investigator's determination. The patient requires a thoracotomy to repair the esophagus and is not amenable for laparoscopic or robotic minimally invasive gastric pull-up (GPU) surgery, due to a medical contraindication
7. All patients must be made aware and must be amenable to a delayed rescue repair surgical procedure in the event the CEI fails to restore a patent durable biologic esophageal conduit
8. The patient/guardian is willing and able to comply with the protocol specified medication regimen and follow-up evaluations
9. The patient/guardian has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Inclusion Criteria Cohort 2:

1. Subject ≥18 years of age
2. The patient has medical conditions requiring esophageal reconstruction, limited to:

   a. Spit Fistula with an upper esophageal ostomy in the neck
3. Patients may require esophageal de-functioning with a resulting cervical spit fistula if they are not candidates for immediate esophageal reconstruction. This may occur for multiple reasons, including being too sick for reconstruction, healing of the airway after tracheo-esophageal fistula repair, requirement for further therapy prior to reconstruction, or recovering from sepsis due to esophageal perforation.
4. The patient must be a surgical candidate for a short segment esophageal reconstruction (< 7cm), a full circumferential segmental esophageal extension in order to have sufficient length to make the anastomosis to the distal thoracic esophagus, to a gastric or to an intestinal interposition conduit that will re-establish oral nutritional intake. i.
5. Patient must be a high-risk candidate for the standard of care treatment of esophageal reconstruction, based upon the investigator's determination. The patient requires a thoracotomy to repair the esophagus following the CEI subdermal extension procedure and is not amenable for laparoscopic or robotic minimally invasive gastric pull-up (GPU) surgery.
6. All patients must be made aware and must be amenable to a delayed rescue repair surgical procedure in the event the CEI fails to mature in the subdermal area prior to mobilization
7. The patient/guardian is willing and able to comply with the protocol- specified medication regimen and follow-up evaluations
8. The patient/guardian has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Exclusion Criteria all cohorts:

1. Subject requires or undergoes an esophageal segmental excision >6 cm in length
2. Esophageal segment extends below the diaphragm or <4 cm below larynx
3. Pre-existing implants/structures adjacent to target surgical location for implant that could cause abrasion of the scaffold/regenerated tissue (e.g., pacemaker lead, vascular clips, vascular grafts).
4. Known clinical contraindication that would obfuscate the use of the covered metallic stent to be used as an adjunct to the procedure
5. Post ablation stricture for Barrett's esophagus treated less than 1 year prior to planned procedure
6. Patient has a comorbidity or contraindication that would preclude any study required procedures including adipose tissue biopsy and esophageal resection surgery. Comorbidities are defined from a subset of the Charlson Comorbidities Index (CCI, Yamashita 2018) scoring system and include:

   1. diabetes mellitus (CCI = 1)
   2. connective tissue disorders (CCI=1)
   3. immune compromised
   4. chemotherapy radiotherapy or chemoradiotherapy (within 60 day clearance)
   5. inability to tolerate major thoracotomy
   6. active infection at the biopsy or thoracotomy incision site
   7. peripheral vascular disease (CCI=1)
   8. all patients with a CCI> 2
7. Life expectancy of less than 1 year
8. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7days prior to index procedure.
9. Has a known untreated neurological, psychological, psychiatric, or other disorder that would interfere with trial endpoints or with cooperation with the requirements of the trial
10. Has a diagnosis of immunodeficiency, receiving cancer therapy including chimeric antigen receptor T cells (CAR-T), receiving systemic steroid therapy (>10 mg prednisone or equivalent daily dose), or any other form of pharmacologic therapy that would inhibit the intended cell growth (e.g., protease inhibitors, immunosuppressants, anti-cytokine therapies) within 30 days prior to index procedure or intended for use during any time after implantation through 12 months post-index procedure.
11. Patient with an infection requiring antibiotic therapy
12. Known allergy to Nitinol (for adjunctive self-expanding covered metallic stent procedure)
13. Current participation in another investigational drug or device study
14. Patient is a prisoner
15. If in the opinion of the investigator, the patient requires pain management (potentially opioid medications) as a result of study participation, the patient is at an unreasonable risk of addiction. This decision may be based upon medical or social history, personal situation, or the expected time course, length, and type of medication use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: The number of patients who develop continuous biologic neo-conduit within the esophagus based on CT/MRI imaging and visual endoscopic evaluation. | Month 3
  The number of patients who develops continuous biologic neo-conduit within the esophagus based on CT/MRI imaging and visual endoscopic evaluation, prior to or at Month 3 visit (Day 77 ±10) following implantation.
All Cohorts: The number of patients who does not develop anastomotic leak or fistula that requires non-endoscopic therapy. | 42 days
  The number of patients who does not develop anastomotic leak or fistula that requires non-endoscopic therapy.
All Cohorts: The number of patients within the first 42 days that do not require a fall back emergency esophagectomy procedure | 42 days
  The number of patients within the first 42 days that do not require a fall back emergency esophagectomy procedure (gastric pull-up, colonic interposition, or other surgical reconstruction).
All Cohorts: Number of participants experiencing death within 30 days of index procedure | Within 30 days
  Number of participants experiencing death within 30 days of index procedure
Cohort 2: The number of patients with maturation of the CEI graft under the dermal layer followed by mobilization and connection to the distal esophagus within the thoracic cavity to form a continuous biologic neo-conduit based on endoscopic evaluation | Month 3
  The number of patients with maturation of the CEI graft under the dermal layer followed by mobilization and connection to the distal esophagus within the thoracic cavity to form a continuous biologic neo-conduit based on endoscopic evaluation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota